CLINICAL TRIAL: NCT03899753
Title: Closure After Total Shoulder Arthroplasty: Subcuticular Closure With 2-Octyl Cyanoacrylate Versus 2-Octyl Cyanoacrylate With A Self-Adhering Mesh (Dermabond Prineo)
Brief Title: Closure After Total Shoulder Arthroplasty: Prineo vs Dermabond
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed by the Einstein IRB
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018-9370
Record Dates: First submitted 2019-02-17; First posted 2019-04-02 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Shoulder Arthritis; Shoulder Arthropathy Associated With Other Conditions
Keywords: prino; total shoulder arthroplasty; wound closure

STUDY DESIGN:
Intervention Model Description: * Prospective Randomized Design
  o After determining a participant's eligibility for inclusion, participant will be randomized to the OCA mesh group or monocryl with dermabond group. After surgery, both groups will be seen at the 2 week, 6 week, and 3 month appointments
Who Masked: Participant, Investigator
Masking Description: Sealed envelop determining which arm the participant is assigned to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 2-Octyl Cyanoacrylate and mesh (Experimental): The wound will be closed with 2-Octyl Cyanoacrylate and a mesh
  Interventions: Device: 2-Octyl Cyanoacrylate and Mesh
- 2-Octyl Cyanoacrylate (Active Comparator): The wound will be closed with just 2-Octyl Cyanoacrylate
  Interventions: Device: 2-Octyl Cyanoacrylate

INTERVENTIONS:
Device: 2-Octyl Cyanoacrylate and Mesh — 2-Octyl Cyanoacrylate and a mesh will be applied to final closure of wounds after undergoing a Total Shoulder Arthroplasty
  Other Names: Prineo
  Arms: 2-Octyl Cyanoacrylate and mesh
Device: 2-Octyl Cyanoacrylate — Incisions will be closed with 2-Octyl Cyanoacrylate after undergoing a Total shoulder arthroplasty
  Other Names: Dermabond
  Arms: 2-Octyl Cyanoacrylate

SUMMARY:
The objective is to compare two types of wound closure after total shoulder arthroplasty to determine which closure is faster, and subsequently if there are different outcomes between the two types of closures.

The objective of this study is to compare two types of wound closure after total shoulder arthroplasty procedures. A single fellowship trained shoulder surgeon will perform all procedures. It is hypothesized that participants who undergo an 2-Octyl Cyanoacrylate (OCA) mesh closure will have a faster closure time, lower cost, non-inferior complication rate, and non-inferior satisfaction scores with respect postoperative follow up and scar appearance.

Participants in the OCA mesh cohort will be compared to participants who have a closure with a running monocryl suture and dermabond. This investigation seeks to determine if OCA closure mesh closure is non-inferior to monocryl suture and dermabond in terms of operative time, cost, complications, and aesthetic appearance.

If the hypothesis is confirmed, this study will suggest that a OCA mesh closure may be used for total shoulder arthroplasty surgeries as an alternative to current conventional closures and may provide a cost benefit.

ELIGIBILITY:
Inclusion Criteria:

* Total shoulder arthroplasty
* Reverse total shoulder arthroplasty
* Age 18-100
* Single Surgeon

Exclusion Criteria:

* Previous shoulder surgery
* Known wound healing complications
* DM, chronic steroid use, vascular insufficiency, morbid obesity (BMI>40), ESRD, family hx of pathologic scars
* Patients on blood thinners (ASA 81mg ok)
* Connective tissue disease
* Allergy to skin adhesive
* Mentally unable to complete questionnaires
* Previous wound over planned incision

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Gruson, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Jack D. Weiler Hospital-Division of Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SH, Wise BL, Zhang Y, Szabo RM. Increasing incidence of shoulder arthroplasty in the United States. J Bone Joint Surg Am. 2011 Dec 21;93(24):2249-54. doi: 10.2106/JBJS.J.01994. PMID 22258770
- [Background] Martin JG, Hollenbeck ST, Janas G, Makar RA, Pabon-Ramos WM, Suhocki PV, Miller MJ, Sopko DR, Smith TP, Kim CY. Randomized Controlled Trial of Octyl Cyanoacrylate Skin Adhesive versus Subcuticular Suture for Skin Closure after Implantable Venous Port Placement. J Vasc Interv Radiol. 2017 Jan;28(1):111-116. doi: 10.1016/j.jvir.2016.08.009. Epub 2016 Nov 9. PMID 27836404
- [Background] Grimaldi L, Cuomo R, Brandi C, Botteri G, Nisi G, D'Aniello C. Octyl-2-cyanoacrylate adhesive for skin closure: eight years experience. In Vivo. 2015 Jan-Feb;29(1):145-8. PMID 25600545
- [Background] Imbuldeniya AM, Rashid A, Murphy JP. A comparison of 2-octyl cyanoacrylate with nylon for wound closure of knee arthroscopy portals. J Wound Care. 2014 Sep;23(9):456-8, 460. doi: 10.12968/jowc.2014.23.9.456. PMID 25284299
- [Background] Freitas-Junior R, Paulinelli RR, Rahal RM, Moreira MA, Oliveira EL, Aiko KF, Approbato MS. The use of 2-octyl cyanoacrylate or nylon suture for skin closure produces similar modifications in scar tissue (an animal model). J Plast Reconstr Aesthet Surg. 2008 Aug;61(8):990-2. doi: 10.1016/j.bjps.2007.11.052. Epub 2008 May 9. No abstract available. PMID 18472319
- [Background] Prince D, Solanki Z, Varughese R, Mastej J, Prince D. Antibacterial effect and proposed mechanism of action of a topical surgical adhesive. Am J Infect Control. 2018 Jan;46(1):26-29. doi: 10.1016/j.ajic.2017.07.008. Epub 2017 Aug 24. PMID 28844382
- [Background] Rushbrook JL, White G, Kidger L, Marsh P, Taggart TF. The antibacterial effect of 2-octyl cyanoacrylate (Dermabond(R)) skin adhesive. J Infect Prev. 2014 Nov;15(6):236-239. doi: 10.1177/1757177414551562. Epub 2014 Nov 30. PMID 28989390
- [Background] Clark JJC, Abildgaard JT, Backes J, Hawkins RJ. Preventing infection in shoulder surgery. J Shoulder Elbow Surg. 2018 Jul;27(7):1333-1341. doi: 10.1016/j.jse.2017.12.028. Epub 2018 Feb 12. PMID 29444755
- [Background] Krebs VE, Elmallah RK, Khlopas A, Chughtai M, Bonutti PM, Roche M, Mont MA. Wound Closure Techniques for Total Knee Arthroplasty: An Evidence-Based Review of the Literature. J Arthroplasty. 2018 Feb;33(2):633-638. doi: 10.1016/j.arth.2017.09.032. Epub 2017 Sep 25. PMID 29066251
- [Background] El-Gazzar Y, Smith DC, Kim SJ, Hirsh DM, Blum Y, Cobelli M, Cohen HW. The use of dermabond(R) as an adjunct to wound closure after total knee arthroplasty: examining immediate post-operative wound drainage. J Arthroplasty. 2013 Apr;28(4):553-6. doi: 10.1016/j.arth.2012.07.038. Epub 2012 Oct 29. PMID 23114193
- [Background] Glennie RA, Korczak A, Naudie DD, Bryant DM, Howard JL. MONOCRYL and DERMABOND vs Staples in Total Hip Arthroplasty Performed Through a Lateral Skin Incision: A Randomized Controlled Trial Using a Patient-Centered Assessment Tool. J Arthroplasty. 2017 Aug;32(8):2431-2435. doi: 10.1016/j.arth.2017.02.042. Epub 2017 Feb 24. PMID 28438450
- [Background] Mudd CD, Boudreau JA, Moed BR. A prospective randomized comparison of two skin closure techniques in acetabular fracture surgery. J Orthop Traumatol. 2014 Sep;15(3):189-94. doi: 10.1007/s10195-013-0282-7. Epub 2013 Dec 31. PMID 24379118
- [Background] Parvizi D, Friedl H, Schintler MV, Rappl T, Laback C, Wiedner M, Vasiljeva A, Kamolz LP, Spendel S. Use of 2-octyl cyanoacrylate together with a self-adhering mesh (Dermabond Prineo) for skin closure following abdominoplasty: an open, prospective, controlled, randomized, clinical study. Aesthetic Plast Surg. 2013 Jun;37(3):529-37. doi: 10.1007/s00266-013-0123-3. Epub 2013 Apr 24. PMID 23613192
- [Background] Richter D, Stoff A, Ramakrishnan V, Exner K, Jernbeck J, Blondeel PN. A comparison of a new skin closure device and intradermal sutures in the closure of full-thickness surgical incisions. Plast Reconstr Surg. 2012 Oct;130(4):843-850. doi: 10.1097/PRS.0b013e318262f237. PMID 23018695
- [Background] Holte AJ, Tofte JN, Dahlberg GJ, Noiseux N. Use of 2-Octyl Cyanoacrylate Adhesive and Polyester Mesh for Wound Closure in Primary Knee Arthroplasty. Orthopedics. 2017 Sep 1;40(5):e784-e787. doi: 10.3928/01477447-20170531-03. Epub 2017 Jun 9. PMID 28598492
- [Background] Sutton N, Schmitz ND, Johnston SS. Economic and clinical comparison of 2-octyl cyanoacrylate/polymer mesh tape with skin staples in total knee replacement. J Wound Care. 2018 Apr 1;27(Sup4):S12-S22. doi: 10.12968/jowc.2018.27.Sup4.S12. PMID 29641342

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled into the study. In the interest of safeguarding the identity of this individual, demographic information is not being disclosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants] — Population: Only 1 participant was enrolled into the study. In the interest of safeguarding the identity of this individual, participant age is not being disclosed.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only 1 participant was enrolled into the study. In the interest of safeguarding the identity of this individual, gender is not being disclosed.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Time for Incision Closure
Description: A stopwatch will be used to measure the time it takes for the incision to be closed. When the surgical implants are in place and irrigation is complete, the surgeon will announce that he will start the closure and a nurse will start the stopwatch to measure how long it takes for the surgeon to close the incision.
Time Frame: During surgery (approximately 40 minutes)
Population: Data was not collected/aggregated and therefore not analyzed.
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cost of Closure
Description: Cost of closure will be assessed by the cost of the time in the operating room and the cost of materials used to close the incision
Time Frame: Immediately post surgery
Population: Data was not collected/aggregated and therefore not analyzed.
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Wound Appearance
Description: The surgeon and participant will fill out the Patient and Observer Scar Assessment Scale (POSAS). This is a survey used to assess the participant and the surgeons opinion of the appearance of the wound. The Patient and Observer Scar Assessment Scale (POSAS) is a questionnaire that was developed to assess scar quality. It consists of two separate six-item scales (Observer Scale and Patient Scale), both of which are scored on a 10-point rating scale. Each questionnaire consists of 7 questions, each graded 1 through 10. The minimum score is 7 (most like normal skin) and the maximum score is 70 (very different from normal skin). The observer is the surgeon. The observer and patient scores can then be added together to determine the collective score.
Time Frame: At each follow up visit up to 3 months after surgery
Population: Data was not collected/aggregated and therefore not analyzed.
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Dehiscence
Description: The wound will be assessed for dehiscence (incision opening) which will be recorded as a "yes or no". A dehiscence is defined as exposure of the underlying subcutaneous fat secondary to failure of the epidermal healing and may be accompanied by persistent wound drainage. It will be assessed by the length of the opening in centimeters and then normalized against the length of the entire incision. Furthermore, the number of wounds that open will be reported
Time Frame: At each follow up visit up to 3 months after surgery
Population: Data was not collected/aggregated and therefore not analyzed.
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Wound Drainage
Description: Dressing for each participant after surgery will be regulated and changed by the surgeon at the first post op visit. Drainage will be measured by outlining the drainage on gauze onto graph paper and measuring the area as previously validated in prior studies
Time Frame: At first post operative visit
Population: Data was not collected/aggregated and therefore not analyzed.
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Superficial Infection
Description: Number of wounds with superficial skin infections will be reported
Time Frame: At each follow up visit up to 3 months after surgery
Population: Data was not collected/aggregated and therefore not analyzed.
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Deep Wound Infection
Description: Number of deep wound infections found will be reported
Time Frame: At each follow up visit up to 3 months after surgery
Population: Data was not collected/aggregated and therefore not analyzed.
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Wounds That Require Post Operative Intervention
Description: Will report the number of wounds that require post operative intervention
Time Frame: At each follow up visit up to 3 months after surgery
Population: Data was not collected/aggregated and therefore not analyzed.
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1-year
Arm/Group | 2-Octyl Cyanoacrylate and Mesh | 2-Octyl Cyanoacrylate
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Only 1 participant was enrolled into the study. In the interest of safeguarding the identity of the individual, demographic information is not being disclosed. Data was not collected/aggregated and therefore not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03899753/Prot_SAP_000.pdf